CLINICAL TRIAL: NCT07215702
Title: A Phase IIa, Randomised, Double-blind, Placebo-controlled, Multicentre Study to Assess the Efficacy, Safety, and Tolerability of AZD4144 in Participants With Sepsis-associated Acute Kidney Injury (SERENIA)
Brief Title: A Study to Investigate the Efficacy, Safety, and Tolerability of AZD4144in Participants With Sepsis-associated Acute Kidney Injury.
Acronym: SERENIA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9440C00004; 2025-522232-13-00 (Registry Identifier: EU CT number); 54675 (Other: CTIS)
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: Sepsis; Acute Kidney Injury; Glomerular Filtration
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, multicentre study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind; Investigators, blinded Sponsor staff, site staff, and participants will remain blinded to each participant's assigned study intervention throughout the course of the study (with the exception of the site pharmacist(s) or designee preparing the IMP and unblinded Monitors/CRAs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (AZD4144) (Experimental): AZD4144 solution for IV infusion
  Interventions: Drug: AZD4144
- Arm 2 (Placebo) (Placebo Comparator): Placebo concentrate for solution for infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4144 — Intravenous solution of AZD4144 will be administered to randomised participants according to the treatment arm to which they have been assigned.
  Arms: Arm 1 (AZD4144)
Drug: Placebo — Intravenous solution of Placebo will be administered to randomised participants according to the treatment arm to which they have been assigned.
  Arms: Arm 2 (Placebo)

SUMMARY:
This study will enroll adults aged 18 to 80 years diagnosed with sepsis due to a suspected or confirmed bacterial infection, within 7 days of being admitted to the hospital, and who have also developed acute kidney injury within 72 hours of the onset of sepsis. Eligible participants will be randomly assigned to receive either AZD4144 or a placebo intravenously once daily for the number of days specified in the CSP. During this Treatment Period, participants will undergo daily safety monitoring, as well as blood and urine sample collection and other assessments. After the Treatment Period, participants will continue to be monitored for safety and other assessments during each additional day they remain hospitalized (if applicable) as well as during up to 2 follow up visits after discharge. The main goal is to compare specific kidney function measurements between those participants receiving AZD4144 and those receiving the placebo.

DETAILED DESCRIPTION:
This is a Phase IIa, randomised, double-blind, placebo-controlled, multicenter study that will be conducted in adult participants (aged 18-80) with sepsis-associated acute kidney injury (SA-AKI). Eligible participants must have sepsis secondary to suspected or confirmed bacterial infection requiring vasopressor or inotrope therapy, and AKI (KDIGO Stage ≥ 1) within a defined time frame of sepsis onset. Participants will be randomised in a 1:1 ratio to receive either intravenous AZD4144 or matching placebo once daily for a fixed treatment period. The study will be comprised of:

* A screening period
* A treatment period, during which participants receive intravenous AZD4144 or placebo daily according to the protocol dosing days.
* A follow-up period that will include daily assessments while still hospitalized and up to two additional outpatient visits at scheduled times after discharge.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 to ≤ 80 years at the time of signing the informed consent.
* Participants who are admitted to an ICU.
* Diagnosis of sepsis according to criteria defined by The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) based on:

  1. Suspected or confirmed bacterial infection AND
  2. Acute increase of mSOFA score of 2 or more excluding renal component (change in score measured to account for participants that may meet mSOFA criteria from pre-existing organ dysfunction before the onset of infection).
* Vasopressor and/or inotrope therapy for sepsis-induced hypotension
* Diagnosis of AKI with modified KDIGO Stage ≥ 1 persisting after initial volume resuscitation (30 mL/kg or as clinically indicated per investigator discretion) defined as: Increase in serum creatinine to ≥ 1.5 × baseline (pre-AKI reference).
* Outpatient pre-AKI reference eGFR ≥ 30 mL/min/1.73 m2 or admission pre-AKI reference eGFR ≥ 45 mL/min/1.73 m2.
* Body weight ≥ 40 kg or ≤ 125 kg.
* Female or male, assigned at birth, inclusive of all gender identities.
* All FOCBP must have a negative pregnancy test at the Screening visit (Visit 1).
* Contraception:

  1. Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods detailed in CSP from the time of first administration of study intervention administration until 100 days after the last dose of study intervention.
  2. FOCBP must not be lactating and must agree to use an approved method of highly effective contraception, as detailed in the CSP from the time of first administration of study intervention until 100 days after last dose of study intervention.
* Capable of giving signed informed consent (participant or LAR)
* Provision of signed and dated written Optional Genomics Initiative Research Information and Consent Form prior to collection of samples for optional genomics initiative research

Exclusion Criteria

* Any clinical evidence which in the investigator's opinion makes it undesirable for the potential participant to enrol in the study.
* Known history of Stage 4 or 5 CKD with documented sustained eGFR < 30 mL/min/1.73 m2 prior to hospital admission.
* No serum creatinine results available within 12 months of admission and an eGFR < 45 mL/min/1.73 m2 at admission.
* Sepsis diagnosed > 7 days after hospital admission (to include from time of outside admission if patient transferred from another healthcare setting).
* AKI attributed to causes other than sepsis, including but not limited to compromised renal perfusion-related causes (surgical complication, acute abdominal aortic aneurysm, dissection, renal artery stenosis, etc), glomerular disease, acute interstitial nephritis, and medication toxicity.
* Evidence of recovery from AKI prior to randomisation defined as:

  1. A reduction of serum creatinine to less than 1.5 times reference serum creatinine in the last available local SoC laboratory result before randomisation or
  2. A > 25% reduction in serum creatinine from peak serum creatinine after volume resuscitation prior to randomisation.
* Expected survival from sepsis < 24 hours.
* Expected survival < 90 days due to chronic or pre-existing medical conditions other than SA-AKI
* Known history of renal transplant or bilateral nephrectomy.
* Permanent incapacitation.
* Active cancer or cancer in remission for less than 2 years.
* Known history of immunodeficiency disease or currently receiving immunosuppressant therapy for non-sepsis related disease.
* Severe burns requiring ICU treatment.
* Sepsis attributed to confirmed or presumed fungal or viral infection at time of Screening.
* Has advanced chronic liver disease, confirmed by a Child-Pugh score of 10-15 (Class C).
* Known history of cerebrovascular accident within the last 90 days.
* Known history of heart failure with reduced ejection fraction with documented ejection fraction ≤ 20% before sepsis diagnosis.
* Known hypersensitivity to iohexol or known history of severe adverse reaction to iodinated contrast media.
* Participants with known medical or psychological condition(s), or who, in the judgement of the investigator, should not participate in the study if they are unlikely to comply with study procedures, restrictions, and requirements.
* Current KRT (eg, continuous haemofiltration and haemodialysis/continuous renal replacement therapy, intermittent haemodialysis, and peritoneal dialysis) or planned KRT at randomisation
* Currently receiving active treatment for malignancy.
* Potential participants will be excluded if they have received a certain class of medication during the weeks before enrollment or are anticipated to require a specific class of medication during the trial duration.

Participants with a known hypersensitivity to AZD4144 or any of the excipients of the product.

* Receipt of another IMP within 30 days, 5 half-lives, or the time frame of expected PD effect from most recent dose, whichever is longest.
* Previous receipt of AZD4144.
* Active or planned treatment of sepsis with an extracorporeal haemoperfusion device.
* Participation in any other concurrent ICU study which could impact participant clinical outcomes and confound results of this study to, including but not limited to volume resuscitation, vasopressor, or mechanical ventilation studies.
* Presence of anuria (≥ 12 hours) at randomisation.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead ECG, at Screening, as judged by the investigator.
* Prolonged QTcF > 470 ms.
* Known history of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* Known history of ST-elevation myocardial infarction or non-ST-elevation myocardial infarction, with or without intervention by percutaneous coronary intervention or coronary artery bypass grafting within the last 90 days.
* Ventricular arrhythmia requiring treatment.
* Known or presumed latent or active tuberculosis.
* Acute pancreatitis with no established source of infection.
* Undergoing extracorporeal membrane oxygenation (ECMO) at randomisation.
* Neutropenia: ANC < 1.5 × 109/L.
* Admitting diagnosis of rhabdomyolysis.
* Admitting diagnosis of trauma with CK > 15000 U/L.
* Presumed nidus of infection in central nervous system.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous randomisation in the present study.
* For females only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
* First dose of IMP unable to be administered within 36 hours of AKI diagnosis.
* Presence of a do-not-resuscitate order.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2027-02-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of 24-hour Creatinine Clearance (CrCl). | During the treatment period.
  The total area under the curve for 24-hour creatinine clearance measured throughout the treatment period.

SECONDARY OUTCOMES:
Days alive and free of KRT. | Through study completion, an average of 30 days.
  The total number of calendar days in which a patient is both alive and not receiving Kidney Replacement Therapy (KRT), such as dialysis.
Days alive and free of modified KDIGO AKI Stage 2 or 3. | Through study completion, an average of 30 days
  The total number of calendar days in which a patient is alive and does not meet criteria for modified KDIGO Acute Kidney Injury (AKI) Stage 2 or 3. The modified KDIGO is a scale measuring AKI severity, ranging from 1 to 3 (most severe).
AUC: Serum Creatinine | During the treatment period.
  The area under the curve for serum creatinine to evaluate changes in renal function.
AUC: Serum Cystatin C | During the treatment period
  The area under the curve for serum cystatin C to evaluate changes in renal function.
AUC: mGFR | During the treatment period.
  The area under the curve for mGFR to evaluate changes in renal function.
Cmax/Cbaseline: Serum creatinine | During the treatment period.
  The ratio of peak serum creatinine to baseline.
Cmax/Cbaseline: Serum cystatin C | During the treatment period.
  The ratio of peak serum Cystatin C to baseline.
AUC: Plasma IL-18 | During the treatment period.
  The area under the curve for plasma interleukin-18 measured as a marker of inflammation.
AUC: Urine IL-18 | During the treatment period.
  The area under the curve for urine interleukin-18 measured as a marker of inflammation.
AUC: Plasma IL-6 | During the treatment period.
  The area under the curve for plasma interleukin-6 measured as a marker of inflammation.
AUC: Urine IL-6 | During the treatment period.
  The area under the curve for urine interleukin-6 measured as a marker of inflammation.
Plasma concentrations of AZD4144 | Through study completion, an average of 30 days
  Measurement of AZD4144 plasma levels to evaluate pharmacokinetics in participants with SA-AKI.
Occurrence of MAKE30 | Through study completion, an average of 30 days
  MAKE30 is defined as the occurrence of any of the following:
  * Decrease from pre-AKI reference eGFR ≥ 25% at Day 30,
  * Initiation of KRT at any time before Day 30,
  * Death from any cause up to Day 30.
Days alive and free of mechanical ventilation | Through study completion, an average of 30 days.
  The total number of calendar days of which a patient is alive and not receiving mechanical ventilation.
Days alive and outside of the ICU | Through study completion, an average of 30 days.
  The total number of calendar days of which a patient is alive and not admitted to the intensive care unit (ICU).
Rehospitalisation | Through study completion, an average of 30 days.
  Occurrence of hospital readmission after initial discharge.
Days alive and free of hospitalisation | Through study completion, an average of 30 days.
  The total number of calendar days of which a patient is alive and not hospitalized.
Days alive and free of vasopressor and/or inotrope | Through study completion, an average of 30 days.
  The total number of calendar days of which a patient is alive and not requiring vasopressor or inotrope support.
AUC mSOFA score | During the treatment period.
  The area under the curve for the modified Sequential Organ Failure Assessment (mSOFA) score to assess organ dysfunction. The modified mSOFA score is a scale to assess organ dysfunction, ranging from 0 (best outcome) to 4 (worst outcome).

CONTACTS AND LOCATIONS:
Locations (58):
- United States (11):
  - Research Site, Tucson, Arizona
  - Research Site, Newport Beach, California
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, The Bronx, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Corvallis, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Salt Lake City, Utah
- Argentina (4):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Rosario
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ottignies
- Canada (2):
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Prague, Czechia
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
- France (5):
  - Research Site, Angers
  - Research Site, La Roche-sur-Yon
  - Research Site, Limoges
  - Research Site, Strasbourg
  - Research Site, Tours
- Germany (6):
  - Research Site, Aachen
  - Research Site, Frankfurt
  - Research Site, Greifswald
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Tatabánya
- Italy (4):
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Jerez de la Frontera
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Kahramanmaraş
  - Research Site, Kocaeli
- United Kingdom (4):
  - Research Site, Brighton
  - Research Site, Guildford
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. ''Yes", indicates that AZ is accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/